CLINICAL TRIAL: NCT05926492
Title: A Prospective, Multicenter, Non-randomized Controlled Clinical Study of Surufatinib Combined With Chemotherapy as Neoadjuvant Treatment in Patients With Osteosarcoma
Brief Title: A Clinical Study of Surufatinib Combined With Chemotherapy as Neoadjuvant Treatment in Osteosarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0425
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-06

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — surufatinib; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surufatinib plus chemotherapy (Experimental): Patients were to receive surufatinib plus chemotherapy every 30 days as neoadjuvant treatment. After receiving 2 cycles of treatment, patients will be evaluated for tumor necrosis rate.
  Interventions: Drug: Surufatinib plus chemotherapy
- Chemotherapy (Active Comparator): Patients were to receive chemotherapy every 30 days as neoadjuvant treatment. After receiving 2 cycles of treatment, patients will be evaluated for tumor necrosis rate.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Surufatinib plus chemotherapy — Surufatinib: (1) for patients aged > 21 years old and ≤70 years old, surufatinib 200 mg, qd, oral, continuous administration; (2) For patients aged ≥2 years and ≤21 years, starting from the low dose of patient BSA (body surface area), Stevenson's formula developed according to the Chinese population was used: BSA = 0.0061H+0.0128W-0.1529 (H: BSA = 0.0061H+0.0128W-0.1529). Height /cm; W: body weight /kg); Chemotherapy : 1) Doxorubicin 60 mg/m2, or liposome doxorubicin 45mg/ m2, day 17; 2) Cisplatin: 100 mg/m2, day 15; 3) Ifosfamide; 2.5g/m2, day 8-12;
  The above drugs were used in turn, and 30 days were regarded as a treatment cycle.
  Other Names: Arm A
  Arms: Surufatinib plus chemotherapy
Drug: Chemotherapy — 1) High-dose methotrexate : 8-12 g/m2 (MTX chemotherapy requires blood drug concentration monitoring), day 1 and 8; 2) Doxorubicin 60 mg/m2 or liposomal doxorubicin 45mg/ m2, day 17; 3) Cisplatin: 100 mg/m2, day 15;4) Ifosfamide; 2.5 g/m2, day 8-12.
  The above drugs were used in turn, and 30 days were regarded as a treatment cycle.
  Other Names: Arm B
  Arms: Chemotherapy

SUMMARY:
This phase II study aims to explore the tumor necrosis rate in osteosarcoma patients treated with a neoadjuvant regimen of surufatinib combined with chemotherapy.

DETAILED DESCRIPTION:
Surufatinib is a potent inhibitor of colony-stimulating factor 1 receptor（CSF-1R）, which shows a promising tumor inhibition effect on sarcoma. This is a prospective, multicenter, controlled phase II study to explore the efficacy and safety of surufatinib combined with chemotherapy in neoadjuvant treatment of osteosarcoma. In this study, 160 patients were enrolled into the following treatment groups with a 1:1 ratio: (1) Surufatinib + chemotherapy group (N=80) (2) control group: chemotherapy group (N=80); A 30-day treatment cycle was performed, the efficacy was evaluated after 2 cycles of neoadjuvant therapy. The primary endpoints were tumor necrosis rate, and secondary endpoints were 1-year progression-free survival (PFS) and drug safety.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood the study and voluntarily signed the informed consent;
2. Age from 2 to 70 years old (inclusive), both male and female;
3. histologically or cytologically confirmed diagnosis of primary bone tumor
4. having at least one measurable lesion (RECIST 1.1);
5. The patient has not been treated before (including any chemotherapy, targeting, immune and other drugs);
6. The functions of major organs and bone marrow are basically normal;
7. ECOG performance status 0 or 1 (PS 0-2 points for amputees);
8. Expected survival ≥12 weeks;
9. Blood test (without blood transfusion within 14 days) 1) Neutrophil absolute value ≥1.5×109/L, platelets ≥100×109/L, hemoglobin concentration ≥9g/dL); 2) Liver function test (aspartate aminotransferase and glutamic aminotransferase ≤2.5×ULN, total bilirubin ≤1.5×ULN; In case of liver metastasis, AST and ALT≤5×ULN); 3) Renal function (serum creatinine ≤1.5×ULN, creatinine clearance (CCr)≥60ml/min);
10. Fertile male or female patients voluntarily used effective contraceptive methods, such as double barrier methods, condoms, oral or injectable contraceptives, intrauterine devices, etc., during the study period and within 6 months of the last study dose. All female patients will be considered fertile unless the female patient has undergone natural menopause, artificial menopause or sterilization (such as hysterectomy, bilateral adnexectomy or radiation of the ovary).

Exclusion Criteria:

1. Patients who have previously received chemotherapy drugs, surufatinib, or other antiangiogenic agents;
2. Received approved or under development systematic anti-tumor therapy within 4 weeks before enrollment, including chemotherapy, radical radiotherapy, biological immunotherapy, targeted therapy, etc.;
3. Received any surgery or invasive treatment or operation (except intravenous catheterization, puncture drainage, etc.) within 4 weeks before enrollment;
4. International Standardized Ratio (INR)> 1.5 or partially activated prothrombin time (APTT) > 1.5×ULN;
5. The investigator identified clinically significant electrolyte abnormalities;
6. The patient currently has hypertension that cannot be controlled by drugs, as follows: systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;
7. Unsatisfactory blood glucose control (FBG > 10 mmol/L);
8. The patient has any current disease or condition that affects the absorption of the drug, or the patient cannot take surufatinib orally;
9. The patient currently has gastrointestinal diseases such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding from unresected tumors, or other conditions determined by researchers that may cause gastrointestinal bleeding or perforation;
10. Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding >30 mL within 3 months , hematemesis, stool, stool blood), hemoptysis ( > 5 mL of fresh blood within 4 weeks) or had a thromboembolic event (including stroke events and/or transient ischemic attacks) within 12 months;
11. Clinically significant cardiovascular disease, including but not limited to the following: acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) Grades for Congestive Heart Failure was > level 2; Ventricular arrhythmias requiring medical treatment; LVEF (Left ventricular Ejection Fraction) < 50%;
12. Have had other malignancies within the past 5 years, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
13. Active or uncontrolled severe infection; 1) Known human immunodeficiency virus (HIV) infection; 2) Known history of clinically significant liver disease, including viral hepatitis [active HBV infection, i.e., HBV DNA positive (> 1×104 copies /mL or > 2000 IU/ml) must be excluded for known hepatitis B virus (HBV) carriers; 3) Known hepatitis C virus infection (HCV) and HCV RNA positive (> 1×103 copies /mL), or other hepatitis, cirrhosis;
14. The patient has current central nervous system (CNS) metastases or previous brain metastases;
15. Patients with persistent toxicity due to any previous antitumor therapy that has not returned to ≤ grade 2, but with alopecia or lymphocytopenia of any grade are admitted to this study;
16. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;
17. Received blood transfusion therapy, blood products and hematopoietic factors, such as albumin and granulocyte colony-stimulating factor (G-CSF), within 14 days before enrollment;
18. Any other medical condition, clinically significant metabolic abnormality, physical abnormality or laboratory abnormality, which, in the investigator's judgment, reasonably suspects that the patient has a medical condition or condition that is not suitable for the use of the investigational drug (such as having seizures and requiring treatment), or which would affect the interpretation of the study results or place the patient at high risk;
19. Urine routine indicated urinary protein ≥2+, and 24-hour urinary protein quantification >1.0g.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Tumor cell necrosis rate (TCNR) | 12 months
  The percentage of patients with tumor cell necrosis > 90% was assessed according to Huvos

SECONDARY OUTCOMES:
1 year Progression-free survival (PFS) rate | 1 year
  The proportion of patients who were free from disease progression or death from any cause within 1 year from enrollment.
All adverse event/Serious adverse event that occurred during the study period according to CTCAE 5.0 | 24 months
  Safety analysis

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China